CLINICAL TRIAL: NCT03595787
Title: Feasibility Study of Tripartite Prehabilitation of Patients With Acute Myeloid Leukaemia and High-risk Myelodysplastic Syndromes During Intensive Chemotherapy Before Allogenic Haematopoietic Stem Cell Transplantation: the COHABILIT Protocol
Brief Title: COaching and Prehabilitation: Faisability Study in Patients With Acute Myeloid Leukemia and Myelodysplastic Syndrome
Acronym: COHABILIT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: COHABILIT-IPC 2017-046
Record Dates: First submitted 2018-07-11; First posted 2018-07-23 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndromes
Keywords: prehabilitation; coaching; nutritional support; physical activity; allogeneic stem cells transplantation
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Motor Activity | interventions — Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prehabilitation program (Experimental): Program based on nutritional support, physical activity program and coaching. Home-based monitoring will be done thanks to connected watches (step counter pedometer) and a connected body fat weight scale
  Interventions: Procedure: Coaching and Habilitation

INTERVENTIONS:
Procedure: Coaching and Habilitation — nutritional support, adapted physical activity and coaching

SUMMARY:
This faisability study aims to evaluate the adhesion of the patient to a multidisciplinary program (adapted physical activity, coaching and nutrition)

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute myeloid leukemia or high-risk myelodysplastic syndrome
* Age between 18 and 70 years
* Eligible for an intensive chemotherapy
* Eligible for allograft
* Able to answer a questionnaire

Exclusion Criteria:

* Diagnosis of acute promyelocytic Leukemia
* Palliative treatment
* Contraindication to moderate physical activity
* Performans status 4, unless it is related to the disease
* Patient who does not understand French
* Patient unable to use a smartphone
* Patient deprived of liberty or placed under the authority of a tutor,
* Patient considered socially or psychologically unable to comply with the treatment and the required medical follow-up.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-04-04 (Actual); Primary Completion 2025-05-04 (Estimated); Study Completion 2025-05-04 (Estimated)

PRIMARY OUTCOMES:
feasibility to the adapted multidisciplinary program | 6 months
  proportion of patients who will complete more than 50% of the APA/coaching sessions prescribed

SECONDARY OUTCOMES:
Evaluate change in functional capacity | 6 months
  Test SPPB
Evaluate changes in upper limb strengt | 6 months
  Prehension strength with handgrip
Evaluate changes in lower limb strength | 6 months
  Quadriceps strength with dynamometer
Evaluate physical activity sessions modalities | 6 months
  Data from connected watch
Evaluate physical activity sessions feasability | 6 months
  Number of sessions not undertaken and reason for refusal
Evaluate positive and negative affect | 6 months
  Outcomes of questionaries : PANAS,
Evaluate life satisfaction | 6 months
  Outcomes of questionaries LSS
Evaluate the level of depression | 6 months
  Outcomes of questionaries HADS
Evaluate the quality of the trainer-trainee relationship | 6 months
  Outcomes of questionaries CART-Q
Evaluate self-efficacy | 6 months
  Outcomes of questionaries Self-efficacy
Evaluate relationship dynamics | 6 months
  Semi-directive interviews
Evaluate QoL | 6 months
  Outcomes of questionaries FACT-Leu
Evaluate the cancer related fatigue | 6 months
  Outcomes of questionaries FACT-Fa
Evaluate correlation between APA coaching sessions undertaken and NRM | 6 months
  Correlation between number of APA sessions and NRM
Evaluate correlation between APA coaching sessions undertaken and survival | 6 months
  Correlation between number of APA sessions and survival rates
Evaluate correlation between APA coaching sessions undertaken and QoL | 6 months
  Correlation between number of APA sessions and Fact-Leu
Evaluate correlation between APA coaching sessions undertaken and fatigue | 6 months
  Correlation between number of APA sessions and Fact-Fa
Evaluate changes in weight | 6 months
  Change in weight (impedancemetry data via connected weighing machine)
Evaluate body mass index | 6 months
  Change in body mass index (BMI= Weight/Height²)
changes in impedancemetry data | 6 months
  Impedaneimetry mesures (connected weighing machine): body mass index variations,
Evaluate muscle mass | 6 months
  Change in muscle mass (impedancemetry data via connected weighing machine)
Evaluate fat mass | 6 months
  Abdominal scan by L3 cross-section: Skeletal Muscle Mass Index (SMI= skeletal muscle mass/height)
Evaluate skeletal muscle mass index (SMI) change in the course of the treatment | 6 months
  Abdominal scan by L3 cross-section: Skeletal Muscle Mass Index (SMI= skeletal muscle mass/height)
Evaluate adherence to nutrition programme | 6 months
  Number of days enteral and parenteral nutrition
Study correlation between variation in weight, BMI, muscle mass, fat mass and SMI on physical capacities, QoL, number of infections, number of days of hospitalisation, patients' outcomes (NRM, survival) and GvHD in allotransplant patients. | 6 months
  Correlation between variation in weight, BMI, muscle mass, fat mass and SMI with NRM, overall survival, number of days of hospitalisation, number of infections documented, QoL, physical capacities and GvHD
Complete remision | 6 months
  Complete remision rate
- Evaluate number of infections documented | 6 months
  number of infections documented
evaluate number of days of hospitalisation | 6 months
  number of days of hospitalisation mesured in nights
evaluate rate of early mortality | 30 days
  rate of premature mortality
evaluate rate of overall mortality | 30 days
  rate of overall mortality
evaluate cause of overall mortality | 6 months
  cause of premature mortality
Evaluate rate of non relapse Mortality (RNM) | 6 months
  Rate of NRM
evaluate overall survival | 6 months
  overal survival rate
evaluate survival without relapse | 6 monts
  survival without relapse rate
evaluate survival without events | 6 monts
  survival without events rate
evaluate number of allotransplant patients | 6 monts
  number of allotransplant patients
evalaute number of patients disqualified for allotransplant | 6 monts
  number of patients with transplant indication disqualified for allotransplant
degree of digestive GVH disease | 6 monts
  GVH disease grade
Evaluation of the severity of digestive GVH disease | 6 monts
  severity of GVH desease

CONTACTS AND LOCATIONS:
Overall Officials: Cécile Bannier Braticevic, MD, Principal Investigator — Institut Paoli-Calmettes
Locations (1):
- Institut Paoli Calmettes, Marseille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Saillard C, Cuvelier S, Villaron-Goetgheluck C, Boher JM, Almeida-Lopez L, Le Corroller AG, Denis P, Rivieccio C, Calvin S, Vey N, Bannier-Braticevic C. Tripartite prehabilitation of patients with acute myeloid leukaemia and high-risk myelodysplastic syndromes during intensive chemotherapy before allogeneic haematopoietic stem cell transplantation (COHABILIT): protocol for an innovating prospective multicentre study. BMJ Open. 2024 Mar 29;14(3):e076321. doi: 10.1136/bmjopen-2023-076321. PMID 38553062